CLINICAL TRIAL: NCT01875887
Title: Application of Surgery Planning Software, Rapid Prototyping Model and Preshaped Titanium Plates in Treatment of Bilateral Maxillofacial Post-traumatic Deformities
Brief Title: Treatment of Bilateral Maxillofacial Post-traumatic Deformities
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Junhui Cui, Principal Investigator, West China Hospital
Other Study IDs: cui_owen
Record Dates: First submitted 2013-06-04; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Therapeutics of Bilateral Maxillofacial Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- treat bilateral maxillofacial deformties: treatment of bilateral maxillofacial post-traumatic deformities
  Interventions: Procedure: rapid prototyping technology

INTERVENTIONS:
Procedure: rapid prototyping technology — Rapid prototyping technology was applied in treatment of bilateral maxillofacial post-traumatic deformities

SUMMARY:
Combined application of surgery planning software and rapid prototyping technology and preshaped titanium plates can effectively promote the accuracy of the diagnosis and treatment of bilateral maxillofacial post traumatic deformities, reduce operation time and improve surgical effect.

DETAILED DESCRIPTION:
All patients underwent preoperative CT scan. Firstly, SurgiCase were used to analyze CT data and design preliminary surgery plans. Secondly, three-dimensions resin skull models were produced by rapid prototyping technology. Model surgeries were performed to determine the location, reduction direction and shift distance of osteotomy. Based on the surgical simulation, the preliminary surgery plans were validated and optimized. Then, the titanium plates and mesh were preshaped on the models. Finally, according to the final surgery plans the operations were performed. The operation time, therapeutic effects and complications were observed. The follow-up periods were 1-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral maxillofacial Post-traumatic Deformities

Exclusion Criteria:

* unilateral maxillofacialPost-traumatic Deformities

Ages: 18 Years to 53 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with Bilateral maxillofacial Post-traumatic Deformities
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-05; Primary Completion 2012-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
improvement in mouth openning | from 1 month to 1year
  The follow-ups showed that the degree of mouth opening of all patients were over 30mm.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, DMD, Study Director — Department of Oral & Maxillofacial Surgery, West China Hospital of Stomatology, Sichuan University
Locations (1):
- West China Hospital of Stomatology, Chengdu, Sichuan, China

REFERENCES:
- See also: The West China Hospital of Stomatology has long been ranked as one of the national top hospitals in China — http://www.hxkq.org/